CLINICAL TRIAL: NCT04989166
Title: Effect of Nano-curcumin Supplementation on Hospital Length of Stay, Clinical Outcomes,and Inflammation Level in Mild and Moderate Acute Pancreatitis.
Brief Title: Effect of Nano-curcumin Supplementation in Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28664
Record Dates: First submitted 2021-07-31; First posted 2021-08-04 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-curcumin (Active Comparator): 80mg of Nano-curcumin daily
  Interventions: Dietary Supplement: Nano-curcumin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Nano-curcumin — Nano-curcumin soft gels
  Arms: Nano-curcumin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of nano-curcumin supplementation on hospital length of stay, clinical outcomes, and inflammation level in mild and moderate acute pancreatitis. 42 eligible patients with mild and moderate acute pancreatitis will randomly assign to consume two soft gels each containing 40 mg of nano-curcumin or placebo (control group) every morning and evening for two weeks. Both groups will also receive the standard medical treatment of acute pancreatitis according to relevant guidelines. Patient's blood samples and clinical outcomes will assess on days 0, 1, 2, 3, 4, and 14 of admission. The two groups will also be compared in terms of adverse events and hospital length of stay. Moreover, the patient's hospital readmission due to pancreatitis will be recorded within 90 days of hospitalization.

DETAILED DESCRIPTION:
The dietary intake of patients will be examined by two non-consecutive 24-hour food recalls at baseline and end of the study. The patient's weight (kg) and Body Mass Index (BMI) will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute pancreatitis by at least two of the three following criteria: 1) a history of acute abdominal pain 2) greater than the threefold elevation of the serum amylase and/or lipase level 3) computed tomographic evidence of acute pancreatitis
* Admission within 72 hours of onset of pain
* Age range of 18-75
* Ability to intake soft gels orally

Exclusion Criteria:

* Severe or critical AP on admission
* Pregnancy or lactation
* A history of allergy to curcumin
* Acute exacerbation of chronic pancreatitis
* Prior antioxidant therapy
* Severe co-morbid illness (liver disease including cirrhosis and hepatitis, Renal failure (Cr Cl < 30 ml/min))
* Active infection
* Active malignancy
* Hyperthyroidism
* Persistent organ failure > 48 hours (according to Marshall score)
* On anticoagulant/ anti platelet medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | through study completion, up to 2 weeks
  calculated from the day of admission until the time of discharge from the hospital.

SECONDARY OUTCOMES:
Overall appetite | days 0, 1, 2, 3, 4, and 14 of admission
  patient's appetite based on visual analogue scale
Abdominal pain intensity | days 0, 1, 2, 3, 4, and 14 of admission
  patient's pain intensity according to verbal numerical rating scale (0-10)
CRP | days 0 and 14 of admission
  Serum level of C-reactive protein
Analgesic medications | days 0, 1, 2, 3, 4, and 14
  daily doses of as-needed analgesics
Hospital readmission | up to 90 days
  Patient's readmission to the hospital after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

REFERENCES:
- [Derived] Chegini M, Sadeghi A, Zaeri F, Zamani M, Hekmatdoost A. Nano-curcumin supplementation in patients with mild and moderate acute pancreatitis: A randomized, placebo-controlled trial. Phytother Res. 2023 Nov;37(11):5279-5288. doi: 10.1002/ptr.7958. Epub 2023 Jul 25. PMID 37490939